CLINICAL TRIAL: NCT02214472
Title: Valoración Objetiva y Tratamiento de la rumiación.
Brief Title: Treatment of Rumination by Biofeedback - a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR(AG)200/2011
Record Dates: First submitted 2014-08-06; First posted 2014-08-12 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Rumination Disorders
Keywords: Rumination síndrome; Regurgitation; Vomiting; Biofeedback; Electromyography; Abdominal accommodation
MeSH Terms: conditions — Rumination Syndrome; Gastroesophageal Reflux; Vomiting | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biofeedback (Experimental): Abdomino-thoracic muscle activity after a challenge meal will be recorded by EMG and the signal will be displayed on a monitor in front of the patients; in the biofeedback group, patients will be instructed to control muscle activity.
  Interventions: Behavioral: Biofeedback
- Placebo medication (Placebo Comparator): Electromyography will be recorded but not shown to the patients. Patients will take a pill of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Behavioral: Biofeedback
  Arms: Biofeedback
Drug: Placebo
  Arms: Placebo medication

SUMMARY:
Rumination syndrome is characterized by effortless recurrent regurgitation of recently ingested food into the mouth, with consequent expulsion or re-chewing and swallowing. In a previous study the investigators showed that rumination is produced by an unperceived, somatic response to food ingestion.

After having identified the key mechanisms of rumination, the investigators developed an original EMG guided biofeedback technique with specific targets for correction, based on EMG-guided control of abdomino-thoracic muscular activity, and in a pilot study the investigators showed the potential effectivity of this treatment. The current aim is to validate this previous uncontrolled observation by a formal placebo-controlled, randomized trial.

DETAILED DESCRIPTION:
Abdomino-thoracic muscle activity after a challenge meal will be recorded by EMG and the signal displayed on a monitor and front in the patients: in the biofeedback group, patients will be instructed to control muscle activity, whereas in the placebo group patients will receive a pill of placebo. In each patient 3 sessions will be performed over a 10-day period. Physiological (muscular activity by EMG) and clinical outcomes (number of rumination events by questionnaires administered daily for 10 days) will be measured before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Rumination syndrome

Exclusion Criteria:

* Relevant organic disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of regurgitation episodes | 28 days

SECONDARY OUTCOMES:
Postprandial abdominal symptoms | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Azpiroz, MD, Principal Investigator — Hospital Universitary vall d'Hebron
Locations (2):
- Spain (2):
  - Fernando Azpiroz, Barcelona, Barcelona
  - University Hospital Vall d'Hebron, Barcelona, Catalonia

REFERENCES:
- [Result] Barba E, Burri E, Accarino A, Malagelada C, Rodriguez-Urrutia A, Soldevilla A, Malagelada JR, Azpiroz F. Biofeedback-guided control of abdominothoracic muscular activity reduces regurgitation episodes in patients with rumination. Clin Gastroenterol Hepatol. 2015 Jan;13(1):100-6.e1. doi: 10.1016/j.cgh.2014.04.018. Epub 2014 Apr 24. PMID 24768808
- [Derived] Barba E, Accarino A, Soldevilla A, Malagelada JR, Azpiroz F. Randomized, Placebo-Controlled Trial of Biofeedback for the Treatment of Rumination. Am J Gastroenterol. 2016 Jul;111(7):1007-13. doi: 10.1038/ajg.2016.197. Epub 2016 May 17. PMID 27185077